CLINICAL TRIAL: NCT05178719
Title: Extension of the TOP 1-study (NCT03901989): Treatment of Osteoporosis by Panaceo, Pear Control Study Assessed Effect on Bone Mineral Density and Bone Turnover of Panaceo Compared to Placebo in Osteoporotic Patients
Brief Title: Treatment of Osteoporosis - TOP 2-5 Clinical Studies (Pear Control)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinic K-center (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, DALIBOR KRPAN, Prof.dr.sc. Dalibor Krpan, prim.dr.med., Polyclinic K-center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOP 002-005-2016
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: The clinical study started in a randomized, double-blinded, controlled study aimed to assess the effect of zeolite-intervention in osteoporotic patients on the bone mineral density and bone turnover in comparison to osteoporotic patients. In the rears 2-5 only receiving the study substance.
  The study TOP 2 started with 81 patients with osteoporosis defined according BMD criteria: T score -2, 5 on the femoral neck, and, or T -2, 5 on L1-L5, who have not been treated before, or in whom privies treatment did not been successful, despite a gender or age.
  Subjects were monitored at the start of the study and at the end of each study year. The surrogate markers of bone status are measured as follows: BMD, changes in levels of osteocalcin and beta-crosslaps CTx assay.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PMA-zeolite (Experimental): All subjects receive the substance 3 times per day in a measuring spoon as powder
  Interventions: Device: PMA-zeolite

INTERVENTIONS:
Device: PMA-zeolite — given for a total period of 4 years

SUMMARY:
Due to the fact that bone mineral density (BMD) is a not enough sensitive parameter for assessment of the bone quality and that the changes in BMD are gradually, extension of the clinical follow up is recommended. On that way the result will be more reliable.

Therefore the protocol "TOP 2-5" is the extension of TOP 1-study with a slight change of the study design. All subjects will be treated with Panaceo. It will be a "pear control", where the patient is control to himself, or herself (each patient from "placebo group (TOP1) can be compared after further years of threatment.

Additionally, extension of the follow up will provide an assessment of the fracture risk in a more reliable manner, which is considered as the most preferably outcome in majority clinical studies of osteoporosis treatment, because it is the most important requirement for the acceptance by the regulatory agencies (FDA, EMA).

DETAILED DESCRIPTION:
Pear control study over 4 supplementation years. Study Population: The study population will consist of patients from a previous study (start: 100 and drop out rate) with osteoporosis defined according BMD (bone mineral density) criteria: T score -2, 5 on the femoral neck, and, or T -2, 5 on L1-L5, who has not been treated before, or in whom privies treatment did not been successful, despite a gender or age. Subjects will receive PMA-zeolite .

Demonstration of efficacy of Panaceo in the treatment of osteoporosis by increasing bone mineral density and reduction of fracture risk.

Demonstration of efficacy of Panaceo in the treatment osteoporosis despite of the gender and cause.

Demonstration of efficacy of Panaceo in the patients who was on drug treatment (bisfosfonates or SERM) more than five years without significant improvement or those who are suspected on the bone turnover over-suppression.

Tolerability Safety (adverse events, vital signs, clinical chemistry)

ELIGIBILITY:
Inclusion Criteria:

* 100 subjects with osteoporosis Among those, as a subgroup, 20 subjects with diabetes type 2 and osteoporosis; The osteoporosis- was diagnosed by standard DXA measurement (BMD T-score: - 2.5 or below )

Exclusion Criteria:

* chronic renal failure, secondary osteoporosis

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Change of BMD (Bone mineral density) | 0-6-12 months for a total period of 4 years
  BMD measurements are used to see how well osteoporosis treatments are working
Fractures and fallings | for a total period of 4 years
  Fracture: evaluation if yes) or no) Falling: Fracture as a consequence OR no fracture OR no fallings reported

SECONDARY OUTCOMES:
Change of Bone remodelling marker Osteocalcin | 0-12 months for a total period of 4 years
  Osteocalcin- parameter of the bone formation rate
Change of Bone remodelling marker Betacross laps | 0-12 months for a total period of 4 years
  Betacross laps - parameter of the bone degradation rate

OTHER OUTCOMES:
Intensity of the musculoskeletal pain measured by VAS | 0-12 months for a total period of 4 years
  the scale based on patient's subjective evaluation at the beginning and at the end of the study
Subjective evaluation of the overall health status | 0-12 months for a total period of 4 years
  upon the end of the study in comparison to the beginning

REFERENCES:
- [Derived] Kraljevic Pavelic S, Saftic Martinovic L, Simovic Medica J, Zuvic M, Perdija Z, Krpan D, Eisenwagen S, Orct T, Pavelic K. Clinical Evaluation of a Defined Zeolite-Clinoptilolite Supplementation Effect on the Selected Blood Parameters of Patients. Front Med (Lausanne). 2022 May 27;9:851782. doi: 10.3389/fmed.2022.851782. eCollection 2022. PMID 35712111